CLINICAL TRIAL: NCT01910922
Title: Learning Mechanisms of Food Preferences in 2-3 y. o. Toddlers in Nurseries
Brief Title: Effect of Learning on Vegetable Acceptance by Toddlers
Acronym: WP23_HabEat
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: habeat_wp2.3; FP7/2007-2010 (Other Grant/Funding Number: 7th european PCRDT (FP7/2007-2010))
Record Dates: First submitted 2011-04-06; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Food Preference
Keywords: vegetable acceptance; vegetable intake; vegetable liking; learning mechanisms; repeated exposure to flavor; flavor learning; replace salt with spice
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Repeated exposure Group (RE): Exposure to basic salsify puree during E1-E8
- Flavour-flavour learning-salt (FFL-S): Exposure to salty salsify puree during E1-E8
- Flavour-flavour learning-nutmeg (FFL-N): Exposure to nutmeg-flavored salsify puree during E1-E8

SUMMARY:
The aim of this study is to understand the formation of food preferences from an early age.

DETAILED DESCRIPTION:
The main purpose of this research is to compare the effectiveness of two mechanisms (mere exposure, flavour-flavour learning) in the short and medium term (up to six months after the learning phase) on 2-3 year-old children's vegetable acceptance. the research is conducted on children aged 2 to 3 years in daycares.

ELIGIBILITY:
Inclusion Criteria:

* children between 2 and 3 years,
* attending daycares
* returned signed consent form parents

Exclusion Criteria:

* children with food allergies or manifestations, chronic disease
* or being preterm (<36 weeks gestational age at birth)

Ages: 17 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 2-3 years olds attending nurseries in Dijon city
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Vegetable intake and liking | baseline = Pre-exposure at one week before the beginning of the experimental manipulation (i.e. exposure phase)
  Measure of salsify and carrot puree intake and liking by toddlers at lunch, at pre-exposure before the exposure phase

OTHER OUTCOMES:
Vegetable intake and liking | exposure period: 4 weeks, twice a week
  Measure of salsify puree intake and liking by toddlers at lunch, during the exposure phase
Vegetable intake and liking | Measure at post-exposure one week after the end of the experimental manipulation (i.e. exposure phase)
  Measure of salsify and carrot puree intake and liking by toddlers at lunch, one week after the exposure phase
Vegetable intake and liking | 1-month follow-up, conducted one month after the end of the experimental manipulation (i.e. exposure phase)
  Measure of salsify intake and liking by toddlers at lunch, at follow-up one month after the exposure phase
Vegetable intake and liking | 3-month follow-up conducted three months after the end of the experimental manipulation (i.e. exposure phase)
  Measure of salsify and carrot puree intake and liking by toddlers at lunch, at follow-up three months after the exposure phase
Vegetable intake and liking | 6-month follow-up conducted six months after the end of the experimental manipulation (i.e. exposure phase)
  Measure of salsify and carrot puree intake and liking by toddlers at lunch, at follow-up six months after the exposure phase

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Nicklaus, PhD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement; Sylvie Issanchou, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- CESG, Dijon, France

REFERENCES:
- See also: European project — http://www.habeat.eu/